CLINICAL TRIAL: NCT03391739
Title: CART-19 Cells For Patients With Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia
Brief Title: CART-19 Cells For R/R B-ALL
Acronym: CCFRRBA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Jianda Hu, Director of the department of Hematology, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART-19-03
Record Dates: First submitted 2017-12-30; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Relapsed/Refractory B-cell ALL
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): CART-19 cells treat
  Interventions: Biological: CART-19 cells

INTERVENTIONS:
Biological: CART-19 cells — CART-19 cells treat

SUMMARY:
There are limited treatment options for relapse/refractory B-cell acute lymphoblastic leukemia(ALL). However,CART-19 cells has emerged as a powerful targeted immunotherapy for highly refractory CD19+ acute lymphoblastic leukemia (ALL). This study aims to assess the safety and toxicity of CART-19 cells to patients with relapse/refractory B-cell ALL.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Aged between 1-60 years
* Patients with relapsed/refractory B-cell ALL
* Cardiac: Left ventricular ejection fraction ≥ 50%
* Adequate renal and hepatic function
* Performance status: Karnofsky ≥ 70%

Exclusion Criteria:

* Pregnant or lactating females.
* Any co-morbidity precluding the administration of CART-19 cells.

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20
Dates: Start 2016-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Leukemia free survival | 1 year

SECONDARY OUTCOMES:
Adverse events that are related to treatment | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China